CLINICAL TRIAL: NCT03231839
Title: Identification of Factors Predicting the Success of a Nutritional Intervention to Decrease the Risk of Type 2 Diabetes
Brief Title: Nutritional Prevention of Diabetes Mellitus Type 2
Acronym: NUPREDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, andreas fritsche, Professor, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UTubingen4
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus; Nutritional and Metabolic Diseases; Liver Fat; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Nutritional and Metabolic Diseases; Fatty Liver; Insulin Resistance | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caloric restriction (control) (Placebo Comparator): daily reduction of caloric intake aimed at 400 kcal/day
  Interventions: Behavioral: Caloric restriction
- No red meat (Active Comparator): daily reduction of caloric intake aimed at 400 kcal/day plus no red meat intake
  Interventions: Behavioral: no red meat
- Increased fiber intake (Active Comparator): daily reduction of caloric intake aimed at 400 kcal/day plus increased fiber intake (aim: 40gr/day)
  Interventions: Behavioral: Increased fiber intake

INTERVENTIONS:
Behavioral: Caloric restriction — After the baseline measurements individuals underwent dietary counseling and had 6 sessions with a dietician (after, 1,4,8,12 16 and 20 weeks).
  Arms: Caloric restriction (control)
Behavioral: no red meat — After the baseline measurements individuals underwent dietary counseling and had 6 sessions with a dietician (after, 1,4,8,12 16 and 20 weeks).
  Arms: No red meat
Behavioral: Increased fiber intake — After the baseline measurements individuals underwent dietary counseling and had 6 sessions with a dietician (after, 1,4,8,12 16 and 20 weeks).
  Arms: Increased fiber intake

SUMMARY:
This study investigates the influence of red meat and fibers on glucose metabolism and body fat composition in subjects at increased risk for type 2 diabetes.

DETAILED DESCRIPTION:
The epidemiologic evidence for increased red meat intake and decreased fiber intake as risk factors for T2D is solid. However, few intervention studies have been performed in order to investigate the role of whole-grain intake or the consumption of red meat in glycemic control and prevention of diabetes, yielding contradicting results. Thus, in order to prove causality, further identify potential underlying mechanisms and be able to improve lifestyle modification programs, we performed a randomized, controlled intervention study over six months. The participants are individuals at increased risk for tyoe 2 diabetes. They were randomised to 3 interventions groups: 1) caloric restriction of 400 kcal/day (control group), 2) caloric restriction plus no red meat consumption 3) caloric restriction and increase in fiber intake. Subjects where thoroughly phenotyped by anthropometric parameters, oral glucose tolerance tests, and MRI measurements of body fat composition and iron content in the liver. In this study, we want to compare the effectiveness of reduced caloric intake only versus reduced caloric intake with an additional modification of diet composition in terms of red meat and fiber consumption.

ELIGIBILITY:
Inclusion Criteria:

Individuals at a high risk for Type 2 diabetes:

* positive family history of type 2 diabetes,
* presence of metabolic syndrome,
* body mass index (BMI) > 27 kg/m2,
* diagnosis of impaired glucose tolerance (IGT)
* previous diagnosis of gestational diabetes diabetes

Exclusion Criteria:

Main exclusion criteria

* diagnosis of type 1 or 2 diabetes mellitus
* BMI >45 kg/m²
* presence of serious illness such as cardiovascular, malignant or psychiatric disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
change in glucose metabolism | baseline and six months
  glucose metabolism measured during the oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Insulin secretion | baseline and six months
  Disposition index (insulin sensitivity (Matsuda) x insulinogenic index (IGI))
liver fat | baseline and six months
  measured by magnetic resonance spectroscopy
liver iron content | baseline and six months
  measured by magnetic resonance imaging
body composition | baseline and six months
  measured by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
Not allowed by ethics committee

REFERENCES:
- [Derived] Willmann C, Heni M, Linder K, Wagner R, Stefan N, Machann J, Schulze MB, Joost HG, Haring HU, Fritsche A. Potential effects of reduced red meat compared with increased fiber intake on glucose metabolism and liver fat content: a randomized and controlled dietary intervention study. Am J Clin Nutr. 2019 Feb 1;109(2):288-296. doi: 10.1093/ajcn/nqy307. PMID 30721948